CLINICAL TRIAL: NCT02400398
Title: A Longitudinal, Single Institution Study Evaluating Weight Stability in Advanced Pancreatic Cancer Patients With Cachexia Who Are Receiving Enteral Feeding
Brief Title: Evaluating Weight Stability of Pancreatic Cancer Cachexia Patients
Acronym: PanCax
Status: Completed | Type: Observational
Sponsor: Andrew Hendifar, MD (Other)
Responsible Party: Sponsor-Investigator, Andrew Hendifar, MD, Assistant Professor of Medicine, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Other Study IDs: IIT2014-03-Hendifar-PNCX1
Record Dates: First submitted 2015-01-12; First posted 2015-03-27 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Pancreatic Neoplasms; Pancreatic Cancer; Cachexia; Weight Loss
MeSH Terms: conditions — Pancreatic Neoplasms; Cachexia; Weight Loss | interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: Yes

GROUPS / COHORTS (1):
- Tube feeding with peptide-base formula: The peptide-based formula (Peptamen) will be administered through a gastrojejunal or jejunal feeding tube and dosing will be calculated using the Mifflin St. Jeor equation. It will be administered for three 28-day cycles.
  Interventions: Other: Tube feeding

INTERVENTIONS:
Other: Tube feeding — Jejunal or gastrojejunal tube feeds will be given as continuous feeds via pump with Peptamen (medical food), at the patient's home, for the duration of the protocol and as directed by the nutritionist.
  Other Names: Enteral feeding; Jejunal tube; Gastrojejunal tube

SUMMARY:
Eligible patients will have a diagnosis of both pancreatic adenocarcinoma and cachexia defined as greater than 5% unintentional weight loss within 6 months prior to screening visit. Patients must be greater than 18 years of age; and have greater than 3 months life expectancy.

This study will observe a standard of care intervention (tube feeding) for potential benefit. Peptamen will be administered through a jejunal or a gastrojejunal feeding tube and dosing will be calculated using the Mifflin St. Jeor equation. It will be administered daily for the duration of the protocol.

DETAILED DESCRIPTION:
In this study, we will prospectively evaluate advanced pancreatic adenocarcinoma patients with cachexia, who are receiving enteral feeding, with a peptide based diet (medical food), through a jejunal or gastrojejunal feeding tube. We plan to collect serum samples routinely and establish a cohort of patients with this clinical syndrome. Our aims are to establish the feasibility and efficacy of enteral nutrition and its relationship to meaningful clinical outcomes. Furthermore, we will assess for a correlation between cachexia, activity, and patient reported outcomes on domains of quality of life in an optional activity tracker sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or locally advanced pancreatic cancer patients (can include new or recurrent diagnosis) referred to SOCCI-CSMC for chemotherapy
* Cachexia defined as greater than 5% unexplained weight loss within 6 months prior to screening visit or consultation with medical oncologist
* Candidate for enteral feeding with Peptamen, a peptide based formula. Must have jejunal or gastrojejunal tube either previously placed or at least prior to Day 1 of study
* Age ≥ 18 years.
* ECOG performance status 0-2
* Greater than or equal to 3 month life expectancy
* Ability to understand and the willingness to sign a written informed consent
* May have received prior anti-cancer treatment, complete or partial resection of primary tumor
* Patients must be ambulatory and have access to a smart phone to participate in the activity tracker sub-study

Exclusion Criteria:

* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Malignant ascites requiring paracenteses
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Bowel obstruction, partial or total
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer patients with cachexia receiving enteral feedings by way of gastrojejunal or jejunal tube.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Weight | Change from baseline at 3 months

SECONDARY OUTCOMES:
Change in lean body mass | Change from baseline at 3 months
  Measured by Dexa Scan
Performance Status (ECOG) | Change from baseline at 3 months
Quality of Life (EORTC QLQ-C30) | Change from baseline at 3 months
Response to nutritional management | Change from baseline at 3 months
  Assessment based on tumor biomarkers during enteral feeding period
Food intake assessment by 24-hour recall | Change from baseline at 3 months
Smell and taste alteration by questionnaire | Change from baseline at 3 months
Muscle strength using hand grip strength dynamometer | Change from baseline at 3 months
Survival | 3 years
Activity - steps taken | Change from baseline at 3 months
  As tracked by Fitbit Charge HR biosensor
Activity - number of stairs | Change from baseline at 3 months
  As tracked by Fitbit Charge HR biosensor
Activity - sleep duration and interruptions | Change from baseline at 3 months
  As tracked by Fitbit Charge HR biosensor
Activity - heart rate | Change from baseline at 3 months
  As tracked by Fitbit Charge HR biosensor
Changes in microbiome analysis | Change from baseline at 3 months
  As measured by stool sample microbiome analysis

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hendifar, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No